CLINICAL TRIAL: NCT00431418
Title: The Effect of Sildenafil in Preterm Infants With Evolving Chronic Lung Disease (SPICE Trial): a Pilot Study
Brief Title: The Effect of Sildenafil in Preterm Infants With Evolving Chronic Lung Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mercy Hospital for Women, Australia (Other)
Responsible Party: Principal Investigator, Dr. Kai Konig, Consultant Neonatologist, Mercy Hospital for Women, Australia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R 06/34
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Active Comparator): Sildenafil oral solution.
  Interventions: Drug: Sildenafil
- 2 (Placebo Comparator): Placebo oral solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — Sildenafil oral solution
  Other Names: Revatio(R)
  Arms: 1
Drug: Placebo — Placebo solution
  Arms: 2

SUMMARY:
The purpose of this pilot study is to investigate in a randomised double-blind trial whether treatment with Sildenafil reduces duration of ventilatory support in preterm infants born at 28 weeks of gestation or less.

ELIGIBILITY:
Inclusion Criteria:

* Newborn babies born <28 weeks of gestation who still need ventilatory support via endotracheal tube or have been re-ventilated at day 7 of life.

Exclusion Criteria:

* Congenital heart defects
* Suspected inborn error of metabolism
* Inhaled Nitric Oxide treatment during assessment

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2010-07 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Length of ventilation | 12 months after completion of study

SECONDARY OUTCOMES:
Bronchopulmonary Dysplasia (BPD) | 12 months after completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Kai König, MD, Principal Investigator — Mercy Hospital for Women; Charles P Barfield, MD, Principal Investigator — Mercy Hospital for Women; Chad C Andersen, MD, Principal Investigator — Mercy Hospital for Women
Locations (1):
- Mercy Hospital for Women, Heidelburg, Victoria, Australia